CLINICAL TRIAL: NCT00213876
Title: Research of Molecular and Metabolic Diagnostic Markers in Oligodendrogliomas A and B Comparatively.
Brief Title: Research of Molecular and Metabolic Markers in Oligodendrogliomas Comparatively to Other Brain Tumours
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Other Study IDs: 3154
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Oligodendrogliomas
Keywords: Brain tumours; oligodendrogliomas; allelotyping; SAGE; Presence of molecular abnormalities statistically linked to survival or response to chemotherapy
MeSH Terms: conditions — Oligodendroglioma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
At present, diagnosis of oligodendroglioma is made on histological and radiographic criteria in the French Mayo-Ste Anne classification. The less frequent grade A oligodendrogliomas are characterized by no vascular contrast on RMN evaluation comparatively to grade B forms. This benign histological subtype relapses in few cases with a more aggressive histology. To determine these relapsed cases at diagnosis, a collection of tumour begun in February 2004. Then, our study was designed to identify diagnostic molecular and metabolic markers that could eventually be used as a signature characterising grade A versus grade B oligodendrogliomas. The molecular analysis will use genomic techniques like allelotyping study, quantitative real-time PCR, gene sequencing , serial analysis of genomic expression and immunohistochemistry, since the metabolic study will be the spectroscopic examination of in vivo tumour. This study will include paediatric and adult patients followed for oligodendrogliomas, medulloblastomas and gliomas to compare the different tumour signatures. All these results will be correlated to survival and clinical features.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric and adult patients (> 1 year of age)
* Patient with oligodendroglioma or medulloblastoma or glioma
* Possibility of 3 year follow-up
* Patient consent obtained

Exclusion Criteria:

-

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with oligodendroglioma or medulloblastoma or glioma
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2004-02; Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natacha Entz-Werle, MD, Principal Investigator — Hopitaux Universitaires de Strasbourg
Locations (1):
- Natacha Entz-Werle, Strasbourg, France